CLINICAL TRIAL: NCT02675738
Title: Reliability of the Preoperative Work-up in a Prospective Series of Patients Submitted to Surgery for Cystic Neoplasms of the Pancreas
Brief Title: Reliability of the Preoperative Work-up in Patients Submitted to Surgery for Cystic Neoplasms of the Pancreas
Acronym: NCP-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Luca Frulloni, MD, PhD, Universita di Verona
Other Study IDs: NCP-1
Record Dates: First submitted 2016-01-06; First posted 2016-02-05 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cystic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: good clinical practice

SUMMARY:
Prospective, observational, cohort study to evaluate the reliability of preoperative work-up of patients submitted to surgery for pancreatic cystic neoplasms, in a tertiary referral center. A comparison between the preoperative diagnostic suspicion and the final pathologic report will be done.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pancreatic cystic neoplasms
* indication to surgery

Exclusion Criteria:

* pregnancy, breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from pancreatic cystic neoplasms candidate to surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of cases with confirmed preoperative diagnosis | Through study completion, on average 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona Hospital Trust, Verona, Italy